CLINICAL TRIAL: NCT04409028
Title: The Effect of Coronal Restoration Type of Endodontic Treated Posterior Teeth on Quality of Life and Satisfaction Patients.
Brief Title: The Effect of Coronal Restoration Type on Satisfaction Patients.
Acronym: OHIP-14
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melek ÇAM (Other)
Collaborators: Okan University (Other)
Responsible Party: Sponsor-Investigator, Melek ÇAM, Assist. Prof., Okan University
Organization: Okan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12122018/100
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Quality of Life
Keywords: OHIP-14; Quality of life; Endodontically treated teeth; Composite resin
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indirect restoration (Active Comparator)
  Interventions: Procedure: Coronal restoration
- direct restoration (Active Comparator)
  Interventions: Procedure: Coronal restoration

INTERVENTIONS:
Procedure: Coronal restoration — A restorative material like composite resin is condensed into the cavity of teeth.

SUMMARY:
This study aimed to evaluate the impacts of coronal restorations of endodontic treated posterior teeth (ETPT) on the satisfaction and quality of patient's life. The patients who were chosen for this purpose were asked to fill in 3 questionnaires.Electronic charts and files of patients who received endodontic treatment in our faculty between 2018 and 2020 were reviewed and chosen. The patients included in the study had been treated by the same endodontist and restorative dental specialist. The coronal restoration of the ETPT had to be either direct composite restoration (DCR) or indirect ceramic restoration (ICR). When the data of patient files and database systems were combined, 76 patients were deemed fit for this study. The patients were contacted by phone to request participation in the study. A rendezvous was created for the patients who agreed to get involved in the study, and those who came to the appointment filled in the questionnaires. Demographics, the semantic differential scale, and the OHIP-14 scores provided data that were entered into Minitab 18 software.

DETAILED DESCRIPTION:
This cross-sectional clinical study was approved by the Ethics Committee of the Istanbul Okan University and conducted both at its Endodontics and Restorative Departments of Dentistry Faculty. A query of the Nucleus database (a patient management software) was performed to identify dental charts of patients who received endodontic treatment between December 2018 and January 2020. We searched only for primary endodontic treatment of vital tooth codes, and then selected the same endodontic specialists' patients. A total of 400 teeth were identified for screening. Next, a specified restorative dentistry specialist's patient searched within these patients, and 150 patients were obtained. The study was completed with 68 participants (n=34 each). Then data and radiographs of patients were checked out for the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients who received only one nonsurgical, single visit primary root canal therapy to one posterior tooth (premolar/molar) which has no periapical lesion and Class I/II coronal restoration, (2) patient's restoration had occlusal function for a minimum of 1 year, (3) patients who were ≥18 years old and no pregnancy or breastfeeding status (4) patients who had good oral hygiene and full dentition (5) patients who were on the American Society of Anesthesiology I and II.

Exclusion Criteria:

* Patients with physical disabilities and communication difficulties, periapical abscess, sinus tract, dental caries were excluded from the study. Patients who had other dental treatments such prosthetic crowns, implants, dental bleaching, filling were not included in the study. Those with open apex teeth were also excluded from the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Quality life of patients | one year
  the scores given by participants to OHIP-14 survey

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided